CLINICAL TRIAL: NCT04783519
Title: Research Evaluating Sleep & Trends for Universal Prevention
Acronym: REST-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00012538; 5R34AA026909-02 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-03-05 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Insomnia; Alcohol Use, Unspecified; Marijuana Use
Keywords: Insomnia; Alcohol Use; Marijuana Use; Young Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcohol Drinking; Marijuana Use | interventions — Ethanol; Mass Screening; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BASICS + SLEEP (Experimental): The BASICS + SLEEP intervention will integrate BASICS feedback and the Motivational Interviewing (MI) process described in the BASICS arm with Brief Behavioral Therapy for Insomnia (BBTI) content and materials. The BASICS + SLEEP intervention will be implemented in 2 sessions of 45-75 minutes and 2 telephone booster sessions. We will follow BBTI procedures, including provision of a physiological rationale for insomnia and the importance of behavioral strategies to regulate sleep; introduction of sleep hygiene; discussion of factors that can impede duration and quality of sleep; introduction of sleep restriction and stimulus control strategies and negotiation of an initial sleep restriction schedule; and follow-up evaluation of success and continued refinement to achieve sleep efficiency goals. Booster contacts serve as opportunities to adjust the sleep restriction schedule, problem-solve challenges, and further build motivation.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia (BBTI); Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS)
- BASICS (Active Comparator): The BASICS condition will meet for 2 sessions of 45-75 minutes. Content depends on the degree to which participants discuss the feedback, have questions, and/or explore behavior change options. Therapists review feedback components with participants, eliciting personally relevant reasons to change as domains are explored. When the participant is ambivalent about change, therapists work with them to explore and resolve that ambivalence. The method is non-confrontational and utilizes exploration of personalized graphic feedback (i.e., frequency, quantity, and peak use alongside perceived and actual norms for alcohol/MJ use) to increase motivation for change by highlighting ways alcohol and/or marijuana use could be incongruent with goals or values. Beliefs, expectations, and motives for use are discussed as are strategies to minimize risks and consequences. Booster sessions address questions and problem-solve challenges that have arisen since the session.
  Interventions: Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS)
- Assessment Only Control (No Intervention): Participants in Assessment Only Control (AOC) condition will complete all assessments (including survey, daily, actigraphy) at the same time as participants in the 2 active interventions. AOC will also attend an in-person meeting to verify identity, provide rationale for daily monitoring, control for time/attention, and participants in all conditions including AOC will receive referrals for community services to address alcohol and MJ use, sleep, and other mental health concerns. No participants will be deprived of services; use of outside services will be tracked to assist with interpretation of outcomes. AOC condition will be offered BASICS + SLEEP after 3-month follow-up.

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia (BBTI) — Brief Behavioral Therapy for Insomnia (BBTI) focuses primarily on stimulus control and sleep restriction as well as sleep hygiene recommendations delivered over 2 in-person sessions and 2 brief telephone boosters and is designed to be implemented by nonspecialists in primary care or other non-clinical settings. The intervention is manualized, and clients utilize sleep diaries and workbook assignments to consolidate recommendations.
  Arms: BASICS + SLEEP
Behavioral: Brief Alcohol Screening and Intervention for College Students (BASICS) — Brief Alcohol Screening and Intervention for College Students (BASICS) is a manualized brief intervention targeting alcohol use and consequences among high risk drinkers and includes both personalized feedback regarding drinking norms, consequences, and motives for drinking, as well as protective behavioral skills for reducing heavy episodic drinking and related consequences. BASICS is delivered in a motivational interviewing (MI) style (Miller & Rollnick, 2002) to enhance intrinsic motivation to change drinking and implement protective behavioral strategies. BASICS has been adapted to target marijuana use and has been adapted for use with a variety of populations.
  Other Names: BASICS
  Arms: BASICS; BASICS + SLEEP

SUMMARY:
This study is designed to develop an integrated intervention to reduce alcohol and marijuana use and consequences and improve sleep among young adults with comorbid heavy episodic drinking, marijuana use, and sleep impairment.

DETAILED DESCRIPTION:
This study is designed to develop an integrated intervention to reduce alcohol and MJ use and consequences and improve sleep among young adults (YA) with comorbid heavy episodic drinking (HED), MJ use, and sleep impairment. HED in YA is an important public health problem, with consequences including accidental injury and death, academic or work problems, unsafe and unwanted sex, and development of alcohol use disorders. Many YA with HED also use MJ, often simultaneously, and experience increased harm as a result. Sleep impairment is common and problematic among YA, identified as the 3rd leading barrier to academic success for students and an important risk factor for mental health problems and suicide in YA. Alcohol use has been linked to impaired sleep in adolescent, YA, college, and older adult populations, with bidirectional causal links between alcohol use and impaired sleep, including negative physiological effects of alcohol on the sleep cycle (e.g., suppression of REM sleep), use of alcohol to promote sleep onset which can both increase alcohol use and resultant sleep impairment, and poor sleep hygiene including delayed and variable sleep-wake timing associated with cyclical patterns of alcohol use during evening and/or weekend social events. Comorbidity of HED and sleep impairment is associated with increased consequences of alcohol use, and exacerbates risk of accidents (including automobile accidents), impaired decision-making, and work and academic difficulties. Similar bidirectional relations exist with MJ use and sleep. Despite risks and consequences, alcohol and MJ prevention programs rarely target sleep directly, and the majority of YA interventions for sleep either focus on sleep hygiene broadly in the absence of specific strategies shown to improve sleep or reduce alcohol or MJ use, or have been relatively intensive interventions with insufficient sample size to truly evaluate impacts on sleep or related comorbid alcohol or MJ use. The current study addresses these gaps through developing and evaluating feasibility and preliminary efficacy of a brief, integrated intervention combining efficacious brief motivational feedback and skills for reducing HED and MJ use and consequences (BASICS) with Brief Behavioral Therapy for Insomnia (SLEEP) shown to improve sleep in other populations. Feasibility and efficacy will be evaluated over a 3-month period, using surveys and daily diaries to assess alcohol, MJ, and sleep at post-intervention and 3- months. Specific aims are: 1) Assess feasibility, acceptability, and preliminary efficacy BASICS + SLEEP in reducing alcohol use and consequences, improving sleep, and weakening daily and lagged (next day) relationships between alcohol and MJ use and sleep impairment; and 2) Use diary data to explore daily and lagged relationships between alcohol use, MJ, sleep impairment, and unique YA contextual factor to further inform prevention of comorbid alcohol use, MJ, and sleep impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24, score on the ISI of 10 or higher, reporting at least one heavy drinking episode in the past two weeks, use of marijuana at least once in the past month

Exclusion Criteria:

* Not meeting the Inclusion Criteria

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, PhD, Principal Investigator — University of Washington
Locations (1):
- The Center for the Study of Health and Risk Behaviors, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troxel WM, Germain A, Buysse DJ. Clinical management of insomnia with brief behavioral treatment (BBTI). Behav Sleep Med. 2012 Oct;10(4):266-79. doi: 10.1080/15402002.2011.607200. PMID 22946736
- [Background] Buysse DJ, Germain A, Moul DE, Franzen PL, Brar LK, Fletcher ME, Begley A, Houck PR, Mazumdar S, Reynolds CF 3rd, Monk TH. Efficacy of brief behavioral treatment for chronic insomnia in older adults. Arch Intern Med. 2011 May 23;171(10):887-95. doi: 10.1001/archinternmed.2010.535. Epub 2011 Jan 24. PMID 21263078
- [Background] Larimer ME, Turner AP, Anderson BK, Fader JS, Kilmer JR, Palmer RS, Cronce JM. Evaluating a brief alcohol intervention with fraternities. J Stud Alcohol. 2001 May;62(3):370-80. doi: 10.15288/jsa.2001.62.370. PMID 11414347
- [Background] Marlatt GA, Baer JS, Kivlahan DR, Dimeff LA, Larimer ME, Quigley LA, Somers JM, Williams E. Screening and brief intervention for high-risk college student drinkers: results from a 2-year follow-up assessment. J Consult Clin Psychol. 1998 Aug;66(4):604-15. doi: 10.1037//0022-006x.66.4.604. PMID 9735576
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N=150, aged 18-24) were recruited in spring 2021 - spring 2022 via online advertising (e.g., Instagram/Facebook, Reddit, TikTok, Craigslist) and from young adults responding to advertising or invitations for other studies in the investigators' lab for which they did not meet criteria, who met initial screening criteria for the study and agreed to future contact. Participants recruited from either source completed additional screening and identity verification prior to enrollment.
Groups:
- BASICS: Brief Alcohol Screening and Intervention for College Students (BASICS) is a manualized brief intervention targeting alcohol use and consequences among high-risk drinkers and includes both personalized feedback regarding drinking norms, consequences, motives, and protective behavioral skills for reducing heavy episodic drinking and consequences. BASICS is delivered in a motivational interviewing (MI) style to enhance intrinsic motivation to change and implement protective behavioral strategies and has been adapted to target marijuana use. The BASICS condition will meet for 2 45-75 min. sessions. Content depends on degree to which participants discuss the feedback, have questions, and/or explore behavior change options. Therapists review feedback components with participants, eliciting personally relevant reasons to change as domains are explored. When the participant is ambivalent about change, therapists work with them to explore and resolve ambivalence. The method is non-confrontational and utilizes exploration of personalized graphic feedback (i.e., frequency, quantity, and peak use alongside perceived and actual norms for alcohol/MJ use) to increase motivation for change by highlighting ways alcohol and/or marijuana use could be incongruent with goals or values. Beliefs, expectations, and motives for use are discussed as are strategies to minimize risks and consequences. Booster sessions address questions and problem-solve challenges that have arisen since the session.
Period: Overall Study
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Started | 49 | 51 | 50
Completed | 38 | 37 | 41
Not Completed | 11 | 14 | 9
Not completed — Withdrawal by Subject | 2 | 7 | 3
Not completed — Lost to Follow-up | 9 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- BASICS + SLEEP: The BASICS + SLEEP intervention integrated BASICS feedback and Motivational Interviewing (MI) for alcohol and marijuana use as described in the BASICS arm with Brief Behavioral Therapy for Insomnia (BBTI). The BASICS + SLEEP intervention was implemented in 2 telehealth sessions of 45-75 minutes and 2 telehealth booster sessions (20-30 mins). Sessions provided rationale for insomnia and importance of behavioral strategies to regulate sleep; introduction of sleep hygiene; discussion of factors (including alcohol and cannabis use) that impede duration and quality of sleep; introduction of sleep restriction and stimulus control strategies and negotiation of an initial sleep restriction schedule and alcohol/cannabis goals; and follow-up evaluation of success and continued refinement to achieve sleep efficiency goals. Booster contacts serve as opportunities to adjust the sleep restriction schedule, problem-solve challenges, and further build motivation. The intervention included personalized feedback depicting both alcohol and cannabis use and perceived norms as well as insomnia symptoms. Feedback also addressed personal maintaining factors for insomnia, sleep hygiene factors, and protective behavioral strategies for both alcohol and cannabis use.
- BASICS: The BASICS condition was conducted via telehealth for 2 sessions of 45-75 minutes and 2 telehealth booster sessions (20-30 minutes). Brief Alcohol Screening and Intervention for College Students (BASICS) is a manualized brief intervention targeting alcohol use and consequences among high-risk drinkers and includes both personalized feedback regarding drinking norms, consequences, and motives for drinking, as well as protective behavioral skills for reducing heavy episodic drinking and related consequences. BASICS is delivered in a motivational interviewing (MI) style (Miller & Rollnick, 2002) to enhance intrinsic motivation to change drinking and implement protective behavioral strategies. BASICS has been adapted to target marijuana use and has been adapted for use with a variety of populations. Both alcohol and cannabis content were integrated in this condition but without specific content to address insomnia symptoms.
- Assessment Only Control: Participants in Assessment Only Control (AOC) condition completed all assessments (including survey, daily, actigraphy) at the same time as participants in the 2 active interventions. AOC also attended an in-person meeting to verify identity, provide rationale for daily monitoring, control for time/attention, and participants in all conditions including AOC received referrals for community services to address alcohol and MJ use, sleep, and other mental health concerns. No participants were deprived of services. AOC condition was offered BASICS + SLEEP after the 3-month follow-up.
- Total: Total of all reporting groups
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control | Total
Number analyzed (Participants) | 49 | 51 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 51 | 50 | 150
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — self-reported age in years at time of screening
  years | 21.37 (1.68) | 21.16 (1.78) | 20.74 (1.60) | 21.09 (1.70)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants were asked "What is your current gender identity?". Response options included: "Man, Woman, Non-binary, Transgender man, Transgender woman, Genderqueer/gender non-conforming, A gender not listed here (please specify), No answer". Responses other than "Man" or "Woman" were collapsed to create a "Non-binary/Gender Diverse" group.
  Participants
    Men | 12 | 19 | 13 | 44
    Women | 31 | 28 | 31 | 90
    Non-binary/Gender Diverse | 6 | 4 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 14 | 45
  Male | 36 | 33 | 36 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 16
  Not Hispanic or Latino | 44 | 45 | 45 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 8 | 8 | 7 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 3 | 1 | 5
  White | 31 | 34 | 29 | 94
  More than one race | 6 | 5 | 9 | 20
  Unknown or Not Reported | 2 | 0 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 50 | 150
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: Score on a scale] — The Insomnia Severity Index is a 7-item measure that assesses the severity of both nighttime and daytime aspects of insomnia. Response options utilized a 5-point Likert scale ranging from 0-4 where "0" reflected low symptom endorsement and "4" reflected high symptom endorsement. Responses across the 7 items are summed to create a Total Score. Total Scores range from 0 to 28.
  Score on a scale | 15.04 (3.78) | 15.22 (3.55) | 15.20 (3.53) | 15.15 (3.59)
Patient-Reported Outcomes Information System Short Form v1.0 Sleep-Related Impairment 8a [Mean (Standard Deviation); unit: T-Score] — The Patient-Reported Outcomes Information System Short Form v1.0 Sleep Related Impairment 8a (8-items) assesses self-reported perceptions of impairment due to sleep problems. Response options range from 1=Not at all to 5=Very much and are summed to create a raw score (range 8-40). Raw scores are transformed to T-scores with a population mean of 50 and a standard deviation (SD) of 10, where higher scores indicate greater impairment due to sleep problems. For example, a T-score of 60 is one SD worse than average, whereas a T-score of 40 is one SD better than average.
  T-Score | 63.72 (5.66) | 63.70 (5.30) | 63.76 (6.76) | 63.73 (5.89)
Quantity/Frequency/Peak Alcohol Use Index (QFP) peak item [Mean (Standard Deviation); unit: Peak number of standard drinks] — The Quantity Frequency Peak Alcohol Use Index was used to assess the peak number of standard drinks consumed on their heaviest drinking occasion over the previous month.
  Peak number of standard drinks | 7.80 (3.03) | 7.69 (2.89) | 8.18 (4.21) | 7.89 (3.41)
Quantity/Frequency/Peak Alcohol Use Index (QFP) quantity item [Mean (Standard Deviation); unit: Standard drinks per occasion] — The Quantity Frequency Peak Alcohol Use Index was used to assess typical drinking quantity using the number of drinks consumed during a typical drinking occasion over the previous month.
  Standard drinks per occasion | 3.53 (1.46) | 4.12 (2.96) | 4.16 (2.71) | 3.94 (2.47)
Quantity/Frequency/Peak Alcohol Use Index (QFP) frequency item [Mean (Standard Deviation); unit: Days per week] — The Quantity Frequency Peak Alcohol Use Index was used to assess the frequency of drinking over a typical week over the previous month. Response options range from 0=I do not drink at all to 7=Every day.
  Days per week | 14.16 (5.94) | 13.62 (5.88) | 13.73 (7.12) | 13.84 (6.27)
Daily Drinking Questionnaire (DDQ) [Mean (Standard Deviation); unit: Standard drinks per week] — The Daily Drinking Questionnaire assesses the typical number of drinks consumed on each day of a typical week over the previous month. Responses were summed to create a total score of overall number of standard drinks consumed over a typical week.
  Standard drinks per week | 10.18 (7.41) | 11.29 (8.41) | 13.5 (14.25) | 11.67 (10.49)
Rutgers Alcohol Problems Index [Mean (Standard Deviation); unit: Score on a scale] — The Rutgers Alcohol Problem Index (23 items) assessed negative consequences related to drinking. Two items were added to assess driving after drinking 2 or more drinks and 4 or more drinks. Response options range from 0=Never to 4=More than 10 times. Responses were summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 100.
  Score on a scale | 10.82 (9.09) | 12.33 (14.94) | 8.88 (11.45) | 10.69 (12.11)
Daily Marijuana Questionnaire [Mean (Standard Deviation); unit: Hours high per week] — The Daily Marijuana Questionnaire was used to assess hours high from cannabis use on each day over a typical week in the past month. Items were summed to create a total score of overall number of hours spent high during a typical week in the previous month.
  Hours high per week | 16.06 (17.95) | 16.47 (16.74) | 15.26 (19.22) | 15.93 (17.87)
Marijuana-Related Consequences [Mean (Standard Deviation); unit: Score on a scale] — Marijuana Consequences were assessed with a 29-item measure assessing consequences related to marijuana use. Response options range from 0=Never to 4=More than 10 times. Scores are summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 116.
  Score on a scale | 31.57 (18.88) | 32.78 (20.71) | 30.80 (15.75) | 31.73 (18.47)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index is a 7-item measure that assesses the severity of both nighttime and daytime aspects of insomnia. Response options utilized a 5-point Likert scale ranging from 0-4 where "0" reflected low symptom endorsement and "4" reflected high symptom endorsement. Responses across the 7 items are summed to create a Total Score. Total Scores range from 0 to 28. Total scores of 0-7=No clinically significant insomnia, 8-14=subthreshold insomnia, 15-21=clinical insomnia (moderate severity), and 22-28=clinical insomnia (severe).
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: Difference in number analyzed by condition are due to differences in follow-up participation rates and/or items skipped by participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Score on a scale
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 8.48 (4.73) | 9.69 (3.24) | 11.31 (3.38)
  3 Month Follow-up: number analyzed (Participants) | 35 | 34 | 41
  3 Month Follow-up | 7.14 (4.61) | 8.97 (5.55) | 9.71 (4.00)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .004, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -0.39, 95% CI 2-sided [-0.650 to -0.127]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .118, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -0.21, 95% CI 2-sided [-.482 to .054]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .003, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -0.41, 95% CI 2-sided [-0.674 to -0.142]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority; p = .240, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -0.16, 95% CI 2-sided [-0.428 to 0.107]

2. Primary Outcome: Patient-Reported Outcomes Information System Short Form v1.0 Sleep-Related Impairment 8a (PROMIS SF8 v1.0 SRI)
Description: The Patient-Reported Outcomes Information System Short Form v1.0 Sleep Related Impairment 8a (8-items) assesses self-reported perceptions of impairment due to sleep problems. Response options range from 1=Not at all to 5=Very much and are summed to create a raw score (range 8-40). Raw scores are transformed to T-scores with a population mean of 50 and a standard deviation (SD) of 10, where higher scores indicate greater impairment due to sleep problems. For example, a T-score of 60 is one SD worse than average, whereas a T-score of 40 is one SD better than average.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
T-Score
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 54.06 (7.85) | 57.31 (6.97) | 58.72 (6.38)
  3 Month Follow-up: number analyzed (Participants) | 35 | 34 | 41
  3 Month Follow-up | 52.66 (7.93) | 56.57 (7.27) | 57.11 (7.71)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .003, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -4.88, 95% CI 2-sided [-8.10 to -1.65]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section. Score on measure (T-score method https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3261577/); Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .308, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -1.71, 95% CI 2-sided [-4.98 to 1.57]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month for BASICS+SLEEP vs. AOC reported in this section. Score on measure (T-score method https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3261577/); Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .007, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -4.52, 95% CI 2-sided [-7.8 to -1.25]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month for BASICS vs. AOC reported in this section. Score on measure (T-score method https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3261577/ ); Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .621, Regression, Linear; Models control for age, sex, race, and ethnicity; beta coefficient = -0.83, 95% CI 2-sided [-4.12 to 2.46]

3. Primary Outcome: Quantity/Frequency/Peak Alcohol Use Index (QFP) Peak Item
Description: The Quantity Frequency Peak Alcohol Use Index was used to assess the peak number of standard drinks consumed on their heaviest drinking occasion over the previous month.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Peak number of standard drinks
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Peak number of standard drinks
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 6.45 (3.15) | 5.92 (2.86) | 8.18 (4.77)
  3 Month Follow-up: number analyzed (Participants) | 35 | 34 | 41
  3 Month Follow-up | 5.06 (2.94) | 4.44 (2.71) | 7.24 (5.08)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .054, Mixed Models Analysis; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.802, 95% CI 2-sided [0.641 to 1.003]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .015, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.750, 95% CI 2-sided [0.600 to 0.946]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .013, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.736, 95% CI 2-sided [0.578 to 0.937]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .001, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.658, 95% CI 2-sided [0.513 to 0.844]

4. Primary Outcome: Quantity/Frequency/Peak Alcohol Use Index (QFP) Quantity Item
Description: The Quantity Frequency Peak Alcohol Use Index was used to assess typical drinking quantity using the number of drinks consumed during a typical drinking occasion over the previous month.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Drinks per occasion
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Drinks per occasion
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 2.93 (1.75) | 2.58 (1.61) | 3.36 (2.05)
  3 Month Follow-up: number analyzed (Participants) | 35 | 32 | 41
  3 Month Follow-up | 2.63 (1.48) | 2.41 (1.79) | 3.61 (2.61)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .960, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Poisson model to address overdispersion (Negative binomial would not converge); count/rate ratio = 0.992, 95% CI 2-sided [0.716 to 1.374]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .152, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.782, 95% CI 2-sided [0.506 to 1.094]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .482, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.887, 95% CI 2-sided [0.634 to 1.240]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .020, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.670, 95% CI 2-sided [0.634 to 1.240]

5. Primary Outcome: Quantity/Frequency/Peak Alcohol Use Index (QFP) Frequency Item
Description: The Quantity Frequency Peak Alcohol Use Index was used to assess the frequency of drinking over a typical week over the previous month. Response options range from 0=I do not drink at all to 7=Every day.
Time Frame: Baseline, 3 Month Follow-up (3 months post-Baseline)
Population: Analyses are using 3 Month Follow-up data.
Measure: Mean (Standard Deviation); unit: Days per week
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 35 | 34 | 41
Days per week | 8.49 (6.75) | 6.79 (4.97) | 9.66 (6.19)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .032, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.724, 95% CI 2-sided [0.540 to 0.973]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p < .001, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.588, 95% CI 2-sided [0.432 to 0.800]

6. Primary Outcome: Daily Drinking Questionnaire (DDQ)
Description: The Daily Drinking Questionnaire assesses the typical number of drinks consumed on each day of a typical week over the previous month. Responses were summed to create a total score of overall number of standard drinks consumed over a typical week.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard drinks per week
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Standard drinks per week
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 6.43 (6.77) | 6.50 (6.67) | 11.05 (9.81)
  3 Month Follow-up: number analyzed (Participants) | 35 | 33 | 41
  3 Month Follow-up | 6.09 (6.12) | 4.48 (4.24) | 10.63 (9.86)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .009, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.699, 95% CI 2-sided [0.535 to 0.914]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .005, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.675, 95% CI 2-sided [0.512 to 0.888]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .013, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.698, 95% CI 2-sided [0.526 to 0.928]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p < .001, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.525, 95% CI 2-sided [0.385 to 0.715]

7. Primary Outcome: Rutgers Alcohol Problems Index
Description: The Rutgers Alcohol Problem Index (23 items) assessed negative consequences related to drinking. Two items were added to assess driving after drinking 2 or more drinks and 4 or more drinks. Response options range from 0=Never to 4=More than 10 times. Responses were summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 100.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Score on a scale
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 6.85 (9.41) | 5.25 (6.71) | 7.64 (6.10)
  3 Month Follow-up: number analyzed (Participants) | 35 | 33 | 41
  3 Month Follow-up | 5.57 (7.05) | 5.27 (9.10) | 6.85 (6.52)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .010, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.598, 95% CI 2-sided [0.404 to 0.885]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .001, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.502, 95% CI 2-sided [0.331 to 0.760]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .002, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.516, 95% CI 2-sided [0.337 to 0.790]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .002, Generalized linear mixed model; [statistical method as in outcome 4, analysis 1]; count/rate ratio = 0.506, 95% CI 2-sided [0.330 to 0.774]

8. Secondary Outcome: Daily Marijuana Questionnaire
Description: The Daily Marijuana Questionnaire was used to assess hours high from cannabis use on each day over a typical week in the past month. Items were summed to create a total score of overall number of hours spent high during a typical week.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours high per week
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 39 | 32 | 40
Hours high per week
  Post Assessment: number analyzed (Participants) | 39 | 32 | 39
  Post Assessment | 7.95 (9.56) | 8.34 (8.80) | 11.21 (19.24)
  3 Month Follow-up: number analyzed (Participants) | 34 | 31 | 40
  3 Month Follow-up | 9.18 (11.89) | 8.26 (11.99) | 11.6 (18.75)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category; p = .003, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.628, 95% CI 2-sided [0.462 to 0.853]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category; p = .073, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = .744, 95% CI 2-sided [0.538 to 1.028]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category; p = .090, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.764, 95% CI 2-sided [0.559 to 1.043]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category; p = .013, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.656, 95% CI 2-sided [0.469 to 0.916]

9. Secondary Outcome: Marijuana-Related Consequences
Description: Marijuana Consequences were assessed with a 29-item measure assessing consequences related to marijuana use. Response options range from 0=Never to 4=More than 10 times. Scores are summed to create a total score of problems experienced in the previous 3 months. Possible scores ranged from 0 to 116.
Time Frame: Baseline, Post-Intervention (7 weeks post-Baseline), 3 Month Follow-up (3 months post-Baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
Number analyzed (Participants) | 40 | 36 | 41
Score on a scale
  Post Assessment: number analyzed (Participants) | 40 | 36 | 39
  Post Assessment | 16.10 (15.86) | 14.97 (14.91) | 18.59 (13.78)
  3 Month Follow-up: number analyzed (Participants) | 35 | 33 | 41
  3 Month Follow-up | 19.71 (15.02) | 18.24 (17.19) | 23.17 (12.69)
Statistical Analysis 1: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .087, Generalized linear mixed model; Model controls for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.753, 95% CI 2-sided [0.546 to 1.041]
Statistical Analysis 2: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to Post Assessment for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .078, Generalized linear mixed model; Model controls for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.739, 95% CI 2-sided [0.528 to 1.034]
Statistical Analysis 3: Comparison: BASICS + SLEEP vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS+SLEEP vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .099, Generalized linear mixed model; Models control for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.773, 95% CI 2-sided [0.569 to 1.050]
Statistical Analysis 4: Comparison: BASICS vs Assessment Only Control; Changes from Baseline to 3 Month Follow-up for BASICS vs. AOC reported in this section; Test type: Superiority — Regression model with TIME × CONDITION Interactions, with AOC as reference category was run using sample of N=150; p = .031, Generalized linear mixed model; Model controls for age, sex, race, and ethnicity. Negative binomial model to address overdispersion; count/rate ratio = 0.704, 95% CI 2-sided [0.512 to 0.969]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial screening and final follow-up for each participant, a period of approximately 7 months.
Description: We used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | BASICS + SLEEP | BASICS | Assessment Only Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/50

LIMITATIONS AND CAVEATS:
All study data were collected during the Covid-19 pandemic, which may have impacted substance use and insomnia symptoms among young adult participants. Additional limitations include relatively small sample size in each condition for this preliminary (pilot feasibility) RCT and slightly higher than anticipated attrition for the 3-month follow-up. All findings are based on self-report of alcohol and cannabis use and sleep symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT04783519/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT04783519/SAP_001.pdf